CLINICAL TRIAL: NCT01038011
Title: Efficacy and Safety of Risedronate (Actonel), a Third Generation Bisphosphonate in Patients With Ankylosing Spondylitis: a Phase 2 Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acto_2003
Record Dates: First submitted 2009-12-15; First posted 2009-12-23 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: drug treatment

SUMMARY:
Randomized, controlled, double-blind, multicenter phase II study comparing risedronate 35mg (ActonelR 35mg weekly tablet) versus placebo in patients with active ankylosing spondylitis (AS) treated with standard first and second-line therapies.

Primary efficacy endpoint: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). The time schedule for performing the BASDAI was at screening, upon inclusion (T0), then after 3, 6 and 12 months or at the time of premature withdrawal in case of drop-out.

secondary endpoints:

* Clinical endpoints: The secondary efficacy measures were the following: Bath Ankylosing Spondylitis Functional Index (BASFI) , Bath Ankylosing Spondylitis Metrology Index (BASMI), ASAS (Assessments in Ankylosing Spondylitis) Working Group core set of domains, Spinal pain VAS, ESR, CRP and the percentage of patients achieving 20% or greater decrease in each of these parameters. These parameters were determined at T0, T3, T6, T12 or at the time of premature withdrawal in case of drop-out. The spinal pain assessed by VAS was also done at screening.
* DEXA: Dual Energy X-Ray-Absorptiometry (DEXA) measurements were performed in all patients upon inclusion (T0) and at the end of the study (T12).
* Biochemical markers: selected biochemical markers of bone metabolism were measured at T0, T3, T6 and T12 or at the time of premature withdrawal in case of drop-out using commercially available kits. Bone formation was assessed by serum bone-specific alkaline phosphatase (BAP) and osteocalcin (OC) levels using commercially available kits. Bone resorption was assessed in serum by the C-terminal telopeptide of type I collagen degradation (Crosslaps R) and urinary N-terminal telopeptide of type I collagen degradation (Osteomark R).
* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: •Male or non-pregnant women (only women who are post menopausal, surgically sterile or practicing a reliable method of contraception may be included) aged 20 years or more

* Meeting the Modified New York diagnostic criteria for AS (Van der Linden S et al., 1984)
* Symptoms of active AS for more than 6 months prior to study entry
* Treated by first-line therapy (NSAIDs) for more than 6 months prior to study entry
* Bath AS Disease Activity Index (BASDAI) score of 4 or greater (Garrett S et al, 1994) and
* Spinal pain of 4 or greater on a 10-cm visual analogue scale despite maximum recommended or tolerated doses of NSAIDs given for a minimum of 1 month prior to study entry

Exclusion criteria: •End-stage AS with diffuse involvement of the spine (complete ankylosis)

* Intraarticular corticosteroid injections or IV infusion with methylprednisolone within the past 2 months prior to study entry. Patients with IA corticosteroid injections of the sacroiliac joints within the past 9 months prior to study entry.
* Severe renal insufficiency: serum creatinine > 25% above the upper limit of normal (>177 umol/l)
* Hypocalcemia
* Major surgery within the past 3 months prior to study entry or planned in the ensuing 12 months
* Orthopaedic surgery within the last 12 months
* Severe infections or comorbidities, or active peptic ulcer disease
* Patients who received bisphosphonates in the past 12 months prior to study entry or patients having known allergies to bisphosphonates.
* Patients treated with anti-osteoporotic drugs (except: Calcium and Vit. D) in the past 12 months prior to study entry.
* Patients unable to remain in an upright position (sitting or standing) during a minimum of 30 minutes
* No written informed consent obtained or inability to collaborate to the study design.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Study Completion 2006-08

PRIMARY OUTCOMES:
BASDAI

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No